CLINICAL TRIAL: NCT07238114
Title: Liver Cirrhosis Patients With Invasive Pulmonary Aspergillosis: in Depth Understanding Clinical Host Risk Factors
Acronym: LIVERIPA
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: S68965; IN-BE-131-7804 (Other Grant/Funding Number: Gilead Sciences)
Record Dates: First submitted 2025-09-09; First posted 2025-11-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Liver Cirrhosis; Viral Pneumonia; Fungal Infection; Invasive Pulmonary Aspergillosis; Intensive Care Medicine
MeSH Terms: conditions — Liver Cirrhosis; Pneumonia, Viral; Mycoses; Invasive Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU patients with liver cirrhosis and IPA: The study population includes patients with confirmed or suspected liver cirrhosis who were admitted to the Medical ICU of UZ Leuven.
  Invasive pulmonary aspergillosis (IPA) is a life-threatening fungal infection, historically seen in severely immunocompromised patients. In recent years, it has also been increasingly recognized in ICU patients without classic immunosuppression, including those with viral pneumonia (e.g., influenza, COVID-19) and those with liver cirrhosis and acute-on-chronic liver failure (ACLF).
- ICU patient with liver cirrhosis without IPA: The study population consists of patients with known or suspected liver cirrhosis who were admitted to the Medical ICU of UZ Leuven.

SUMMARY:
Invasive pulmonary aspergillosis (IPA) is a life-threatening fungal infection of the respiratory system, caused by a specific fungus called Aspergillus species. It is already known that patients with a weakened immune system are at higher risk of developing this disease. Recently, it has also been shown that patients with viral pneumonia (such as influenza or COVID-19) and patients with liver cirrhosis who are admitted to the intensive care unit are also vulnerable to this infection.

This study aims to better define the epidemiology, clinical risk factors, outcomes, and treatment of IPA in ACLF patients admitted to the ICU. By combining clinical data with histological findings from autopsies, the study seeks to improve diagnostic accuracy, risk prediction, and timely initiation of antifungal therapy.

ELIGIBILITY:
Inclusion Criteria:

* All adults (≥ 18 years old)
* Acute-on-Chronic liver failure
* Respiratory distress
* Admission to the Medical Intensive Care Unit of University Hospitals of Leuven

Exclusion Criteria:

* Patients < 18 years
* Respiratory distress not being the primary reason for ICU admission
* Patients with influenza or COVID-19
* Recent history of invasive pulmonary aspergilosis and/or invasive candidiasis (<1 month before ICU admission) and/or active treatment for IPA and/or invasive candidiasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with known or suspected liver cirrhosis who were admitted to the Medical ICU of UZ Leuven.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
IPA incidence | From the date of ICU admission until ICU discharge, approximately 7 days
  The incidence of proven invasive pulmonary aspergillosis (IPA) in critically ill cirrhotic patients will be assessed. Routinely used biochemical and microbiological tests (such as galactomannan and Aspergillus PCR) will be performed on blood and BAL samples stored in the biobank to identify affected patients.
Identifying whether ACLF is an independent risk factor for IPA in EORTC-negative critically ill patients | From the date of ICU admission until ICU discharge, approximately 7 days
  The occurrence of IPA will be compared between an ACLF EORTC-negative cohort and a non-ACLF cohort

SECONDARY OUTCOMES:
Clinical characteristics of IPA | From the date of ICU admission until ICU discharge, approximately 7 days
  Baseline characteristics, organ failures, organ support, outcome parameters
Radiological characteristics of IPA | From the date of ICU admission until ICU discharge, approximately 7 days
  Chest CT
Mycological characteristics of IPA | From the date of ICU admission until ICU discharge, approximately 7 days
  Galactomannan testing, Aspergillus PCR, mycological culture
Impact of IPA on length of ICU stay | From the date of ICU admission until ICU discharge, approximately 7 days
Impact of IPA on length of hospital stay | From the date of ICU admission until hospital discharge, approximately 36 days
Impact of IPA on mortality | From ICU admission until 90 days post-admission
Impact of IPA on liver transplant eligibility | From the date of ICU admission until ICU discharge, approximately 7 days
Impact of IPA on liver transplant delisting | From the date of ICU admission until ICU discharge, approximately 7 days
Histological characteristics of IPA using tissue staining | Through study completion, an average of 3 years
  Histological characteristics of IPA in critically ill cirrhotic patients will be analyzed. Additional histological staining (e.g., Grocott stain) will be performed to detect fungal hyphae.
Histological characteristics of IPA using microbiological testing | Through study completion, an average of 3 years
  Histological characteristics of IPA in critically ill cirrhotic patients will be analyzed. Additional microbiological testing (e.g., Aspergillus PCR) will be performed to detect fungal hyphae.
Correlation of pre-mortem data with post-mortem lung tissue findings | Through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Joost Wauters, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium